CLINICAL TRIAL: NCT06924112
Title: Exercise-induced Hypoalgesia Following Blood Flow Restriction in Rotator Cuff Repair Rehabilitation: a Randomized Crossover Clinical Trial
Brief Title: Blood Flow Restriction Exercise-induced Hypoalgesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, José Casaña Granell, Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P-5.2025
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Rotator Cuff Injury; Rotator Cuff Tear; Rotator Cuff Repair
Keywords: blood flow restriction therapy; blood flow restriction training; exercise-induced hypoalgesia
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Opaque sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isometric exercises with BFR (Intervention A) (Experimental): Participants with arthroscopic rotator cuff repair will undergo to a physical therapy session using three isometric exercises with BFR
  Interventions: Other: Isometric exercises; Device: Isometric exercises with BFR
- Isometric exercises alone (Intervention B) (Active Comparator): Participants with arthroscopic rotator cuff repair will undergo to a physical therapy session using three isometric exercises without BFR
  Interventions: Other: Isometric exercises

INTERVENTIONS:
Other: Isometric exercises — The three isometric exercises were performed without the addition of BFR following the best evidence recommendations. Each exercise was performed for 10 repetitions, with isometric contraction of 15 seconds followed by a rest period of 15 seconds, intensity with a load at 20-25% of the maximal voluntary isometric contraction (MVIC), rest period after each exercise of 2 minutes, and pain level below 5 on the verbal Numeric Pain Rating Scale (NPRS).
Device: Isometric exercises with BFR — Participants will perform three isometric exercises with BFR. An auto-regulated portable BFRT SmartCuffs® 3.0 Pro system with a 17-inch long and 5-inch-wide cuff (Smart Tools Plus, United States), placed on the most proximal part of the arm, will be used. The session will begin with a maximal occlusion test to personalize the occlusion pressure to the participant. The limb occlusion pressure (LOP) will be set at 60% of the maximum occlusion pressure. Each exercise was performed for 10 repetitions, with isometric contraction of 15 seconds followed by a rest period of 15 seconds, intensity with a load at 20-25% of the MVIC, rest period after each exercise of 2 minutes with cuff deflated (reperfusion), and pain level below 5 on the NPRS.
  Arms: Isometric exercises with BFR (Intervention A)

SUMMARY:
The goal of this crossover randomized clinical trial is to compare the acute effect on exercise-induced hypoalgesia (EIH) between isometric exercise with blood flow restriction (BFR) and isometric exercise alone in adults undergoing arthroscopic rotator cuff repair. It is presumed that the addition of BFR to isometric exercises induces a greater effect in EIH.

Patients who agree to participate in this research will be randomly assigned to two intervention sequences (AB or BA), where intervention A (experimental) corresponds to isometric exercises with BFR, and intervention B (control) corresponds to isometric exercises alone. For one week, each participant attended two sessions, separated by a 72-hours wash-out period. The primary variables will be the pressure pain threshold (PPT) and conditioned pain modulation (CPM). Secondary variables will be the pain intensity and distribution, kinesiophobia, upper extremity disability, and quality of life. Results will be measured before intervention (T1, pre-intervention), immediate after intervention (T2, post-intervention 1) and 10 minutes after intervention (T3, post-intervention 2).

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-65 years.
* Symptomatic degenerative rotator cuff tear diagnosed by magnetic resonance imaging.
* Undergoing arthroscopic rotator cuff repair
* Be able to read and understand Spanish.

Exclusion Criteria:

* Massive irreparable RC tears, concomitant fracture, labral or nerve injury.
* Suspicion of developing/diagnosis a frozen shoulder.
* Revision surgery after RC repair.
* Previous corticosteroid injection (< 1 year).
* Recent surgery (< 1 year) in the contralateral shoulder.
* A history of deep venous thrombosis/pulmonary embolism.
* Peripheral vascular disease, thrombophilia or clotting disorders.
* Severe or uncontrolled hypertension, or any comorbid condition that prevents participants from complete the intervention.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) | Pre-intervention (T1), inmediate post-intervention (T2) and 10 minutes post-intervention (T3)
  Pressure pain threshold will be taken bilaterally on the deltoid muscle and the upper trapezius muscle using a Wagner FPX25 pressure algometer (kg/cm2/sec)
Condicionated pain modulation (CPM) | Pre-intervention (T1), inmediate post-intervention (T2) and 10 minutes post-intervention (T3)
  Condicionated pain modulation will be measured with a conditioning stimulus of inmersion of the hand contralateral to the operated shoulder in cold water (10°C). The bilateral deltoid and trapezius muscles before and after the conditioning stimulus will be measured using a Wagner FPX25 pressure algometer (kg/cm2/sec)

SECONDARY OUTCOMES:
Pain intensity and distribution | Pre-intervention (T1), inmediate post-intervention (T2) and 10 minutes post-intervention (T3)
  Visual Analogue Scale (0 to 10 centimeters) and pain distribution map (number of areas)
Kinesiophobia | Pre-intervention (T1), inmediate post-intervention (T2) and 10 minutes post-intervention (T3)
  Tampa Scale of Kinesiophobia (11 to 44 points)
Self-reported upper extremity disability | Pre-intervention (T1), inmediate post-intervention (T2) and 10 minutes post-intervention (T3)
  Shoulder Pain Disability Index (0 to 100%)
Self-reported quality of life | Pre-intervention (T1), inmediate post-intervention (T2) and 10 minutes post-intervention (T3)
  Western Ontario Rotator Cuff Index (0 to 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Ponce-Fuentes, MSc, Principal Investigator — Universidad Mayor; Jose Casaña, PhD, Study Director — University of Valencia; Joaquin Calatayud, PhD, Study Director — University of Valencia; Filip Struyf, PhD, Study Director — Universiteit Antwerpen
Locations (1):
- Clínica RedSalud Mayor, Temuco, Cautín, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. J Appl Physiol (1985). 2020 Apr 1;128(4):914-924. doi: 10.1152/japplphysiol.00768.2019. Epub 2020 Feb 27. PMID 32105522
- [Background] Kuppens K, Struyf F, Nijs J, Cras P, Fransen E, Hermans L, Meeus M, Roussel N. Exercise- and Stress-Induced Hypoalgesia in Musicians with and without Shoulder Pain: A Randomized Controlled Crossover Study. Pain Physician. 2016 Feb;19(2):59-68. PMID 26815250
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Ogrezeanu DC, Lopez-Bueno L, Sanchis-Sanchez E, Suso-Marti L, Lopez-Bueno R, Nunez-Cortes R, Cruz-Montecinos C, Perez-Alenda S, Casana J, Gargallo P, Calatayud J. Exercise-induced hypoalgesia with end-stage knee osteoarthritis during different blood flow restriction levels: Sham-controlled crossover study. PM R. 2023 Dec;15(12):1565-1573. doi: 10.1002/pmrj.13076. Epub 2023 Dec 8. PMID 37796567
- [Background] Korakakis V, Whiteley R, Epameinontidis K. Blood Flow Restriction induces hypoalgesia in recreationally active adult male anterior knee pain patients allowing therapeutic exercise loading. Phys Ther Sport. 2018 Jul;32:235-243. doi: 10.1016/j.ptsp.2018.05.021. Epub 2018 May 31. PMID 29879638
- [Background] Rice D, Nijs J, Kosek E, Wideman T, Hasenbring MI, Koltyn K, Graven-Nielsen T, Polli A. Exercise-Induced Hypoalgesia in Pain-Free and Chronic Pain Populations: State of the Art and Future Directions. J Pain. 2019 Nov;20(11):1249-1266. doi: 10.1016/j.jpain.2019.03.005. Epub 2019 Mar 21. PMID 30904519
- [Background] Vaegter HB, Jones MD. Exercise-induced hypoalgesia after acute and regular exercise: experimental and clinical manifestations and possible mechanisms in individuals with and without pain. Pain Rep. 2020 Sep 23;5(5):e823. doi: 10.1097/PR9.0000000000000823. eCollection 2020 Sep-Oct. PMID 33062901
- [Background] Wewege MA, Jones MD. Exercise-Induced Hypoalgesia in Healthy Individuals and People With Chronic Musculoskeletal Pain: A Systematic Review and Meta-Analysis. J Pain. 2021 Jan;22(1):21-31. doi: 10.1016/j.jpain.2020.04.003. Epub 2020 Jun 26. PMID 32599154
- [Background] Kjaer BH, Magnusson SP, Henriksen M, Warming S, Boyle E, Krogsgaard MR, Al-Hamdani A, Juul-Kristensen B. Effects of 12 Weeks of Progressive Early Active Exercise Therapy After Surgical Rotator Cuff Repair: 12 Weeks and 1-Year Results From the CUT-N-MOVE Randomized Controlled Trial. Am J Sports Med. 2021 Feb;49(2):321-331. doi: 10.1177/0363546520983823. Epub 2021 Jan 20. PMID 33471547